CLINICAL TRIAL: NCT03472066
Title: Measurement of the Cervix During Pregnancy According to Age of Conization
Acronym: MesCon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0021
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Cervix; Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- a group of women who have been conized: Previous conization
  Interventions: Other: Previous conization
- control group with asymptomatic patients: on routine second trim no previous conization
  Interventions: Other: no previous conization

INTERVENTIONS:
Other: Previous conization — a group of women who have been conized,
  Groups: a group of women who have been conized
Other: no previous conization — group with asymptomatic patients on routine second trimester echography
  Groups: control group with asymptomatic patients

SUMMARY:
Treatment of precancerous lesions of the cervix by conization has been shown to increase the risk of premature delivery and premature rupture of the membranes. It has now been clearly established that the cervix is a growing organ during adolescence and early adulthood, It has been hypothetized that cervical conization during the growth phase reduced its growth potential, and induced shorter cervix during the upcoming pregnancy. No studies have been conducted investigating the age at which conization no longer had an impact on cervical size during pregnancy. This will help to identify the age at conisation below which patients will be identified as being at risk event, and thus offer increased monitoring and possibly prophylactic management by programmed strapping. We propose to measure the length of the cervix of pregnant patients who have benefited from conization, which is currently recommended by the Collège National des Gynécologues Obstetriciens Français .In addition, the investigators will use a control group consisting of non-con conical, parity-matched pregnant patients in whom a cervical measurement will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred since January 2008 with pregnancy between 2008 and 2017
2. Pregnancy after conisation
3. Cervix size between 21 and 24 SA before any obstetric event
4. Control group: parity matching, asymptomatic patients

Exclusion Criteria:

1. Threat of late miscarriage,
2. Premature rupture of membranes before cervical echography,
3. Other pregnancies after study of 1st pregnancy after conisation,
4. No measurement of the conization specimen,
5. Lost to follow-up,
6. Age <18
7. Twin Pregnancies
8. Patient under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Including 84 evaluable patients for the primary endpoint would show a Pearson correlation of at least 0.3 between cervical size and age at conization. These calculations were carried out with a 5% risk of first bilateral species and 80% power. Taking into account the risk of incomplete data, we plan to include 90 patients. A control group of 90 patients will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-07-19 (Estimated); Study Completion 2019-08-19 (Estimated)

PRIMARY OUTCOMES:
The main objective is to study the correlation between the size of the cervix and the age at conization. age at conization | 1 day
  Cervix length Measured during the second semester echography

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France